CLINICAL TRIAL: NCT00229502
Title: Comparison of the Cognitive Effects of Three Immunomodulatory Drugs in Relapsing-Remitting Multiple Sclerosis: A Longitudinal Study
Brief Title: Cognitive Effects of Immunomodulatory Drugs in MS
Status: Completed | Type: Observational
Sponsor: Sharon Lynch, MD (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor-Investigator, Sharon Lynch, MD, Professor and Director of MS Center, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 10066
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Subjects receiving Avonex
- 2: Subjects receiving Rebif
- 3: Subjects receiving Copaxone
- 4: Healthy controls

SUMMARY:
The purpose of this study is to examine and compare changes in the specific thinking skills of patients with RRMS who are receiving treatment with one of three immunomodulatory medications (Avonex, Copaxone, or Rebif).

DETAILED DESCRIPTION:
In addition this study will compare the patients' personal view of how they are doing, any changes in physical disability, and the frequency and severity of relapses over the three year period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS for at least one year,
* Currently on one of three immunomodulatory drugs (Avonex, Copaxone, or Rebif),
* Visual Acuity is 20/50 or better,
* patient has four color vision,
* Must have at least a high school education

Exclusion Criteria:

* History of head injury, drug/alcohol abuse, and/or psychiatric problems, -current diagnosis of a severe or lifethreatening disease other than MS,
* currently taking immunosuppressant medication,
* resides greater than 200 miles from the study site

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Multiple sclerosis clinic
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon G Lynch, MD, Principal Investigator — University of Kansas Medical Center; Douglas R Denney, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States